CLINICAL TRIAL: NCT03652935
Title: Mindfulness Based Stress Reduction for Psycho-Immune Dysregulation
Brief Title: Mindfulness, Breast Cancer and Psycho-Immune Dysregulation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Loyola University (Other)
Responsible Party: Principal Investigator, Linda Janusek, Professor, Loyola University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 200101
Record Dates: First submitted 2018-08-26; First posted 2018-08-29 (Actual); Last update posted 2018-08-29 (Actual); Status verified 2018-08

CONDITIONS: Breast Cancer
Keywords: Breast cancer, mindfulness, immune, stress
MeSH Terms: conditions — Breast Neoplasms | interventions — Mindfulness-Based Stress Reduction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mindfulness Based Stress Reduction (Experimental): The Mindfulness Based Stress Reduction (MBSR) program consists of an 8-week (2.5 hr/wk) program with a 6-hour silent mindful practice retreat after the fifth week. A licensed clinical psychologist, certified as an MBSR instructor, will provide instruction to all groups. Mindfulness will be taught using breath awareness, sitting and walking meditation, and mindful yoga. Participants will be given a standardized session-by-session program workbook containing weekly objectives and assignments, as well as two practice recordings and the book, Full Catastrophe Living (Kabat-Zinn, J, 1990).
  Interventions: Behavioral: Mindfulness Based Stress Reduction
- Health Education Series (Active Comparator): The active comparator condition consists of an 8-week educational series, administered in group-format, and matched in duration and frequency to the MBSR program. Session topics include: 1) Understanding Breast Cancer and Risks for Breast Cancer, 2) Breast Cancer Treatment, 3) Communicating Effectively with your Health Care Providers; Keeping your Medical Records, 4) Genetic Testing and Cancer, 5) Nutrition and Cancer, (6) Cooking Demonstration, 7) Bone Health, and 8) Image and Cancer (American Cancer Society - Look Good, Feel Better). The program content and objectives were reviewed by four content experts (oncology clinicians) and two breast cancer survivors.
  Interventions: Other: Health Education Series

INTERVENTIONS:
Behavioral: Mindfulness Based Stress Reduction
  Arms: Mindfulness Based Stress Reduction
Other: Health Education Series — This is an active comparator condition that consists of 8 weekly classes related to health.
  Arms: Health Education Series

SUMMARY:
The purpose of this study is to evaluate the benefits of a Mindfulness Based Stress Reduction (MBSR) program for psycho-immune dysregulation in women newly diagnosed with breast cancer compared to women with breast cancer completing an attention control condition (health education classes). Women will be randomized to either the MBSR or health education classes. They will complete psychometric instruments evaluating psychological outcomes and will provide blood samples for immune outcomes. They will also provide saliva samples for cortisol diurnal rhythm determination. Measures will be done longitudinally pre and post MBSR or health education program. It is hypothesized that MBSR participants will exhibit improved psychological and immunological outcomes over time, as compared to women randomized to the health education classes.

DETAILED DESCRIPTION:
The Mindfulness-Based Stress Reduction (MBSR) program is designed to cultivate conscious awareness (i.e., mindfulness) of one's experience in a non-judgmental or accepting manner (Kabat-Zinn, et al., 1990). Mindfulness programs may facilitate recovery from cancer. However, most prior mindfulness investigations for women with breast cancer focused on cancer survivors, well beyond the acute period of cancer diagnosis and treatment. Moreover, few of these studies evaluated immune measures with relevance to cancer.

Women diagnosed with early stage breast cancer (Stages 0, 1, 2, and 3) will be enrolled. Eligible women will be identified after completion of their breast surgery and when surgical pathology reports are available. Women will complete psychometric instruments and study questionnaires. They will provide blood for immune measures and saliva for cortisol diurnal rhythm. Measures will be done at five separate time points. These are pre-, mid-, and completion of either the MBSR or the attention control program, as well as at 1- and 6-months post-program. Demographic information and information about health behaviors will be collected by self-report. Wrist actigraphy for an additional assessment of sleep quality will be done in an exploratory manner. Hierarchical linear modeling will be used to compute multilevel model for change, based on full maximum likelihood estimation (Raudenbush, S. W., and A. S. Bryk. 2002). Hierarchical linear modeling will be applied to examine intra-individual and inter-individual differences in initial status (baseline) and trajectories of change over time.

ELIGIBILITY:
Inclusion Criteria:

* Women
* Early Stage Breast Cancer

Exclusion Criteria:

* Prior training in MBSR,
* Recurrent breast cancer,
* Metastatic breast cancer,
* Other cancers (except basal cell carcinoma),
* Immune-based disease,
* Psychoses,
* Cognitive dysfunction,
* Unable to read or write English,
* History of substance abuse,
* Use of immune-altering medications

Ages: 28 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 192 (Actual)
Dates: Start 2008-09-15 (Actual); Primary Completion 2013-12-16 (Actual); Study Completion 2013-12-16 (Actual)

PRIMARY OUTCOMES:
Change in Natural Killer Cell Activity | Change from baseline NKCA to 36 weeks.
  Natural killer cell lytic activity (NKCA) against tumor targets will be assessed ex vivo using participant peripheral blood mononuclear cells (PBMC) in a standard chromium release assay, as we described previously (Witek-Janusek, L. et al., 2007).
Change in Cytokine Levels | Change from baseline cytokine level to 36 weeks.
  Plasma levels of cytokines, Interleukin 6 (IL-6) and Tumor Necrosis Factor (TNF) alpha and PBMC cytokine production of these cytokines and interferon (IFN) gamma will be determined. Measurement of individual cytokines will be by quantitative sandwich enzyme immunoassay (R & D Systems, Minneapolis, MN), as we described previously (Witek-Janusek, L. et al., 2007; Witek-Janusek, et al., 2008).
Change in Perceived Stress | Change from baseline perceived stress level to 36 weeks.
  The construct, perceived stress, will be measured using the Perceived Stress Scale (Cohen, S. et al., 1983). The Perceived Stress Scale is a 10-item instrument that assesses the degree to which life experiences are appraised as uncontrollable. Individual items are summed, with scores ranging from 0 (minimum) to 40 (maximum); higher scores indicate higher perceived stress.
Change in Depression | Change from baseline depression level to 36 weeks.
  The construct, depression, will be measured using the Center for Epidemiologic Studies - Depression scale. This is a 20-item measure that asks individuals to rate how often over the past week they experienced symptoms associated with depression. Individual items are summed with scores ranging from 0 (minimum) to 60 (maximum); higher scores indicate greater depressive symptoms (Radloff, LS, 1977).
Change in Fatigue | Change from baseline fatigue level to 36 weeks.
  The construct, fatigue, refers to a subjective sense of tiredness. Fatigue will be measured using the Multidimensional Fatigue Symptom Inventory-Short Form, which consists of 30 items that assess the extent of fatigue experienced by the respondent. Individual items are summed with scores ranging from -24 to 96. Higher score indicates greater fatigue (Stein, KD, et al., 2004).
Change in Sleep | Change from baseline sleep quality level to 36 weeks.
  The construct, sleep quality, will be measured using the Pittsburgh Sleep Quality Index, which consists of 19 items that measure a person's perception of their sleep quality. An overall score is calculated by summing items. Scores range from 0 (minimum) to 21 (maximum), where lower scores denote a better sleep quality (Buysse, DJ, et al., 1989).

SECONDARY OUTCOMES:
Change in Cortisol | Change from baseline cortisol level to 36 weeks.
  Cortisol diurnal rhythm is determined by repeated measure of salivary cortisol (Kirschbaum, C and Hellhammer, DH. 1994). This allows frequent non-invasive sampling under everyday conditions. Subjects will collect saliva samples upon awakening (within 15 minutes of awakening), and at 1200, 1700, and 2200 hr on 2 consecutive days. Centrifuged samples will be frozen and assayed in duplicate using immunoassay kits (Salimetrics™), which measure biologically active (non-protein bound) cortisol.
Change in Quality of Life in Cancer | Change from baseline quality of life level to 36 weeks.
  The construct, quality of life, will be measured using the Quality of Life Index Cancer Version III. Quality of life refers to "a person's sense of well-being that stems from satisfaction or dissatisfaction with the areas of life that are important to him/her." Items are summed to provide global quality of life, with score ranging from 0 (minimum) to 30 (maximum); higher scores indicate better quality of life (Ferrans, CE, 1990).
Change in Social Support | Change from baseline social support level to 36 weeks.
  The construct of social support refers to the extent to which a person's social relationships provide support. Social support will be measured using the 24-item Social Provisions scale, which measures the degree of perceived social support. Responses to items are summed and scores range from 24 to 96;a higher score indicates a greater degree of perceived support (Cutrona CE and Russell DW,1987).
Change in Coping | Change from baseline to 36 weeks.
  The construct of coping with cancer will be measured using the Jalowiec Coping Scale. The Jalowiec Coping Scale is a 60 item self-report measure assessing efficacy of coping behaviors. The JCS allows for the respondent to identify which coping behaviors he/she uses and to then rate the effectiveness of that coping behavior. A score of coping effectiveness is calculated. Scores can theoretically range between 0 and 180, with higher scores indicating greater use of coping behaviors (Jalowiec A, et al., 1984).
Change in Wrist Actigraphy Measure of Sleep Quality | Change from baseline actigraphy to 36 weeks.
  Wrist Actigraphy will be used as a measure of sleep quality (Morgenthaler, T. et al. 2007). Women will be given an Actiwatch (Respironics) and asked to wear the Actiwatch for 6 days (non-dominate wrist). Actiwatch software will be used to calculate a composite of sleep quality.

CONTACTS AND LOCATIONS:
Overall Officials: Linda Janusek, PhD, Principal Investigator — Loyola University Chicago

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Morgenthaler T, Alessi C, Friedman L, Owens J, Kapur V, Boehlecke B, Brown T, Chesson A Jr, Coleman J, Lee-Chiong T, Pancer J, Swick TJ; Standards of Practice Committee; American Academy of Sleep Medicine. Practice parameters for the use of actigraphy in the assessment of sleep and sleep disorders: an update for 2007. Sleep. 2007 Apr;30(4):519-29. doi: 10.1093/sleep/30.4.519. PMID 17520797
- [Background] Buysse DJ, Reynolds CF 3rd, Monk TH, Berman SR, Kupfer DJ. The Pittsburgh Sleep Quality Index: a new instrument for psychiatric practice and research. Psychiatry Res. 1989 May;28(2):193-213. doi: 10.1016/0165-1781(89)90047-4. PMID 2748771
- [Background] Cohen S, Kamarck T, Mermelstein R. A global measure of perceived stress. J Health Soc Behav. 1983 Dec;24(4):385-96. No abstract available. PMID 6668417
- [Background] Cutrona CE and Russell DW. 1987. The provisions of social relationships and adaptation to stress. Advances in Personal Relationships. 1:37-6.
- [Background] Ferrans CE. Development of a quality of life index for patients with cancer. Oncol Nurs Forum. 1990 May-Jun;17(3 Suppl):15-9; discussion 20-1. PMID 2342979
- [Background] Jalowiec A, Murphy SP, Powers MJ. Psychometric assessment of the Jalowiec Coping Scale. Nurs Res. 1984 May-Jun;33(3):157-61. PMID 6563533
- [Background] Kabat-Zinn, J. 1990. Full Catastrophe Living. Delacorte, New York.
- [Background] Kirschbaum C, Hellhammer DH. Salivary cortisol in psychoneuroendocrine research: recent developments and applications. Psychoneuroendocrinology. 1994;19(4):313-33. doi: 10.1016/0306-4530(94)90013-2. PMID 8047637
- [Background] Radloff, LS 1977. The CES-D Scale: A self-report depression scale for research in the general population. Applied Psychological Measurement 1:385-401. doi.org/10.1177/014662167700100306
- [Background] Raudenbush, SW and Bryk, AS. 2002. Hierarchical Linear Models: Applications and Data Analysis Methods, 2 ed. Sage, Thousand Oaks, CA.
- [Background] Stein KD, Jacobsen PB, Blanchard CM, Thors C. Further validation of the multidimensional fatigue symptom inventory-short form. J Pain Symptom Manage. 2004 Jan;27(1):14-23. doi: 10.1016/j.jpainsymman.2003.06.003. PMID 14711465
- [Background] Witek-Janusek L, Gabram S, Mathews HL. Psychologic stress, reduced NK cell activity, and cytokine dysregulation in women experiencing diagnostic breast biopsy. Psychoneuroendocrinology. 2007 Jan;32(1):22-35. doi: 10.1016/j.psyneuen.2006.09.011. Epub 2006 Nov 7. PMID 17092654
- [Background] Witek-Janusek L, Albuquerque K, Chroniak KR, Chroniak C, Durazo-Arvizu R, Mathews HL. Effect of mindfulness based stress reduction on immune function, quality of life and coping in women newly diagnosed with early stage breast cancer. Brain Behav Immun. 2008 Aug;22(6):969-81. doi: 10.1016/j.bbi.2008.01.012. Epub 2008 Mar 21. PMID 18359186